CLINICAL TRIAL: NCT04704453
Title: Phase II Randomized Controlled Study Aiming to Evaluate the Interest of Qutenza in Patients With Head and Neck Cancer in Remission and With Sequelae Neuropathic Pain.
Brief Title: Study to Evaluate the Interest of Qutenza in Patients With Head and Neck Cancer in Remission and With Sequelae Neuropathic Pain.
Acronym: TEC-ORL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20 VADS 04
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer
Keywords: Neuropathic Pain; Capsaicin patch; Amitriptyline
MeSH Terms: conditions — Head and Neck Neoplasms; Neuralgia | interventions — Capsaicin; Amitriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (A): capsaicin patch (Experimental)
  Interventions: Drug: Capsaïcin patch (Qutenza®)
- Standard arm (B): amitriptyline (Other)
  Interventions: Drug: Amitriptyline (Laroxyl®)

INTERVENTIONS:
Drug: Capsaïcin patch (Qutenza®) — Treatment by application of capsaicin 8% (Qutenza®) patches 3 months apart (Month 1, Month 4 and Month 7).
  Arms: Experimental arm (A): capsaicin patch
Drug: Amitriptyline (Laroxyl®) — Treatment by amitriptyline (oral solution 40mg/ml), for 9 months at the recommended dose of 25 mg to 75 mg daily.
  Arms: Standard arm (B): amitriptyline

SUMMARY:
This study aims to compare the analgesic activity of capsaicin patch 8% applications at 3 months interval each on the cervico-facial area versus a reference neuropathic treatment with amitriptyline in patients with head and neck cancer in remission and with sequelae neuropathic pain.

In this phase II trial, patients will be assigned in one of the two treatment arms:

* Arm A (Experimental arm): Capsaïcin patch (Qutenza®)
* Arm B (standard arm): Amitriptyline (Laroxyl®)

  130 patients will be included and will be followed during 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. ORL cancer in remission: absence of clinical or radiological signs of progression at least 3 months after specific treatments.
3. Pain of the cervico-facial sphere persisting for more than 3 months after surgical and/or radiotherapy treatment.
4. Peripheral neuropathic character of pain objectified to a score ≥ 4/10 on the DN4 questionnaire.
5. Pain whose average intensity over the last 24 hours is assessed on the numerical scale as ≥ 2/10.
6. Postmenopausal patient or patient who agrees to use effective contraception for the duration of treatment and for a minimum of 15 days after the end of the treatment period. Non-menopausal patients must have a negative pregnancy test prior to inclusion in the study.
7. Patient affiliated to a Social Health Insurance in France.
8. Patient who signed informed consent prior to inclusion in the study and prior to any specific study procedures.

Exclusion Criteria:

1. ORL cancer in progression.
2. Other concomitant neoplasia (progressive or not).
3. Central etiology of pain.
4. Pain whose average intensity over the last 24 hours is assessed on the numerical scale as < 2/10.
5. Allergy to any of the components of the capsaicin patch.
6. Capsaicin patch not applicable to the area to be treated despite the precautions described in the protocol because of its proximity to mucous membranes or eyelids.
7. Contraindication to amitriptyline treatment.
8. Patient with an unhealed skin lesion on the area to be treated.
9. Previous treatment with capsaicin or amitriptyline.
10. Topical treatment of the painful area used for more than 21 days before inclusion.
11. Ongoing opioid treatment > 80mg/day oral morphine equivalent.
12. Uncontrolled high blood pressure or cardiovascular history (infarction, stroke, pulmonary embolism) less than 3 months ago.
13. Patient included in another interventional therapeutic trial.
14. Pregnant or breastfeeding patient.
15. Any psychological, family, geographical or sociological condition that prevents compliance with the medical follow-up and/or procedures of the study protocol.
16. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
The rate of patients with a decrease in average pain over the last 24 hours by 2 points at 9 months compared to inclusion. | 9 months for each patient
  Pain will be assessed using a numerical scale from 0 to 10.

SECONDARY OUTCOMES:
Neuropathic pain according to the Neuropathic Pain Symptom Inventory (NPSI) questionnaire. | 9 months for each patient
Adverse events of the drugs evaluated using the NCI-CTC AE V5. | 9 months for each patient
Quality of life evaluated according to the Quality of Life Questionnaire-Core 30 (QLQ-C30). | 9 months for each patient

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - INSTITUT DE CANCEROLOGIE DE L'OUEST (ICO) Site Angers, Angers
  - Institut Sainte-Catherine, Avignon
  - Hôpital Saint-Joseph, Marseille
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse

REFERENCES:
- [Derived] Boden A, Lusque A, Lodin S, Bourgouin M, Mauries V, Moreau C, Fabre A, Mounier M, Poublanc M, Caunes-Hilary N, Filleron T. Study protocol of the TEC-ORL clinical trial: a randomized comparative phase II trial investigating the analgesic activity of capsaicin vs Laroxyl in head and neck Cancer survivors presenting with neuropathic pain sequelae. BMC Cancer. 2022 Dec 5;22(1):1260. doi: 10.1186/s12885-022-10348-2. PMID 36471253